CLINICAL TRIAL: NCT00213564
Title: Gene Expression Profiling in PBMCs as a Tool for Prediction of Infliximab Responsiveness in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2002/061/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: response to infliximab associated with methotrexate

SUMMARY:
The objective of the study is to identify and validate predictive markers of infliximab responsiveness in RA patients by 2 approaches: i) measuring biochemical, immunological and bone markers in sera because of their involvement in pathogenic mechanisms; ii) identifying gene-expression signatures in PBMCs by the transcriptomic analysis.

Patients with active RA (ACR criteria) were given i.v. 3 mg/kg infliximab associated with metotrexate at weeks 0, 2, 6, and every 8th week. Infliximab efficacy was evaluated at week 14, using the EULAR response criteria.

1. Just before the starting of infliximab treatment, the following parameters were measured in the sera: i) immunological tests: rheumatoid factor (IgA, IgG, IgM), anti-CCP, autoAb recognizing the 27 C-terminal fragment (ACAST-C27) and domain I (ACAST-DI) of calpastatin, anti-G6PI, anti a-enolase, anti-keratin and anti-perinuclear factor; ii) biochemical markers: CRP, MMP-1, MMP-3, TIMP-1, TIMP-2; markers of bone resorption: pyridinolin, deoxypyridinolin, osteoprotegerin, sRANKL, COMP. The predictive value of each parameter for a response/non-response to infliximab was analysed using Fischer's exact, Mann-Whitney and Chi2 tests.
2. A blood sample was collected just before the onset of infliximab treatment and total RNAs were extracted from the peripheral blood mononuclear cells. The [33P] radiolabeled mRNAs were hybridized (duplicate or triplicate) over a set of 10.000 human cDNA probes spotted at a high density on nylon membranes. Data were normalized and filtered to allow the comparison between RNA samples. Statistical analyses were performed with the R software and hierarchical clustering was performed with the Cluster and Tree View softwares.

ELIGIBILITY:
Inclusion Criteria:

* Is age 18 years old or older Satisfies the 1987 American College of Rheumatology revised criteria for Rheumatoid arthritis Has active disease at the time of randomization as indicated by a DAS28> 5.1 Has a disease at least refractory to DMARDs whose methotrexate or leflunomide Is capable of understanding and signing an informed consent form Agrees to use a medically accepted form of contraception during the study

Exclusion Criteria:

* Is pregnant or breast-feeding or without Has significant concurrent medical diseases including cancer or a history of cancer within 5 years of entering the study, uncompensated congestive heart failure, significant active infection or any underlying diseases that could predispose subjects to infections (whose tuberculosis) Has allergy to infliximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-04; Primary Completion 2004-05 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Le Loët, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de Rouen - Hôpitaux de Rouen, Rouen, France